CLINICAL TRIAL: NCT02599207
Title: Assessment of the Safety of Allogeneic Umbilical Cord Blood Infusions in Children With Cerebral Palsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joanne Kurtzberg, MD (Other)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00065043
Record Dates: First submitted 2015-11-02; First posted 2015-11-06 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Matched related umbilical cord blood (Experimental): Six subjects will receive an infusion of HLA matched sibling umbilical cord blood cells.
  Interventions: Biological: sibling umbilical cord blood
- Mismatched related umbilical cord blood (Experimental): Nine subjects will receive an infusion of HLA-mismatched (≥3/6 match) or matched sibling umbilical cord blood cells.
  Interventions: Biological: sibling umbilical cord blood

INTERVENTIONS:
Biological: sibling umbilical cord blood — All subjects will receive a single infusion of allogeneic sibling cord blood. The first six subjects will receive cord blood cells from an HLA-matched sibling. The following 9 subjects will receive cord blood cells from an HLA-mismatched (≥3/6 match) or matched sibling. Six of the 15 subjects must be treated with haplo-identical sibling CB. Duration of study participation will be six months from the time of CB infusion.

SUMMARY:
This study is a single site, phase I, prospective study of the safety of intravenous sibling cord blood infusion in 15 children ages 1-6 years with Cerebral Palsy (CP). All subjects will be treated with sibling cord blood cells. The first six will receive cord blood cells from an HLA-matched sibling. The following nine subjects will receive cord blood cells from an HLA-mismatched (≥3/6 match) or matched sibling. The duration of study participation will be six months from the time of the cord blood infusion.

DETAILED DESCRIPTION:
This study is a phase I, prospective, open-label trial designed to assess the safety of a single allogeneic sibling cord blood infusion in young children with cerebral palsy. Children ages one to six years with uncomplicated cerebral palsy and an available HLA matched or haploidentical, qualified, sibling cord blood unit will be eligible to participate. All participants will receive a single intravenous infusion of allogeneic sibling cord blood. All participants will have an initial clinical evaluation to verify the diagnosis of cerebral palsy and determine eligibility. The main endpoint is safety, for which acute infusion reactions as well as incidence of infections and graft versus host disease will be assessed. Functional outcome measures, described below, will be assessed at baseline and six months post sibling cord blood infusion and described.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥12 months and ≤ 6 years at the time of CB infusion.
2. Diagnosis: Cerebral palsy with diplegia, hemiplegia, or quadriplegia.
3. Performance status:

   * Bilateral cerebral palsy (diplegia or quadraplegia):

   Gross Motor Function Classification Score levels II - IV, or Gross Motor Function Classification Score level I, age ≥ 2 years
   * Hemiplegia: Gross Motor Function Classification Score levels II - IV or minimal functional capabilities in the affected upper extremity. A subject classified as GMFCS level I with significant upper extremity impairment will be eligible if the affected upper extremity is used as an assist only.
4. Review of brain imaging (obtained as standard of care prior to study entry) does not suggest a genetic condition or brain malformation.
5. Suitably matched sibling donor CB unit (see section 6.2 for matching details) available at a private or public cord blood bank with a minimum total nucleated cell dose of ≥ 2.5 x 107 cells/kilogram.
6. Legal authorized representative consent.

Exclusion Criteria:

1. Available qualified autologous cord blood unit
2. Autism and autistic spectrum disorders without motor disability.
3. Hypsarrhythmia.
4. Intractable seizures causing epileptic encephalopathy.
5. Evidence of a progressive neurologic disease.
6. Has an active, uncontrolled systemic infection or documentation of HIV+ status.
7. Known genetic disease or phenotypic evidence of a genetic disease on physical exam.
8. Concurrent genetic or acquired disease or comorbidity(ies) that could require a future allogeneic stem cell transplant.
9. Requires ventilatory support, including home ventilator, CPAP, BiPAP, or supplemental oxygen.
10. Impaired renal or liver function as determined by serum creatinine >1.5mg/dL and/or total bilirubin >1.3mg/dL except in patients with known Gilbert's disease.
11. Possible immunosuppression, defined as WBC <3,000 cells/mL or absolute lymphocyte count (ALC) below normal for age with abnormal T-cell subsets.
12. Patient's medical condition does not permit safe travel.
13. Previously received any form of cellular therapy.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Assessment for infusion reactions, infections, graft versus host disease or any other adverse events | 6 months
  The primary endpoint of this study is safety which will be evaluated by assessing the incidence of acute infusion reactions, infections, graft versus host disease.

SECONDARY OUTCOMES:
Assessment for improvement in gross motor function | 6 months
  Assessment of improvement in gross motor function using validated tools.
Assessment for improvement in fine motor function | 6 months
  Assessment of fine motor function using validated tools.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke University; Jessica Sun, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States